CLINICAL TRIAL: NCT01455181
Title: A 6-Month Open-label Study Investigating the Safety and Tolerability of NPSP558, a Recombinant Human Parathyroid Hormone (rhPTH [1-84]), for the Treatment of Adults With Hypoparathyroidism - A Clinical Extension Study
Brief Title: A Study to Investigate the Safety and Tolerability of NPSP558, for the Treatment of Adults With Hypoparathyroidism - A Clinical Extension Study in Hungary
Acronym: REPEAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAR-C10-009; 2011-001265-40 (EudraCT Number)
Record Dates: First submitted 2011-09-15; First posted 2011-10-19 (Estimated); Results first posted 2015-03-06 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Hypoparathyroidism
Keywords: PTH 1-84; Hypoparathyroidism; NPSP558; Parathyroid Hormone 1-84
MeSH Terms: conditions — Hypoparathyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NPSP558 (Experimental)
  Interventions: Drug: NPSP558

INTERVENTIONS:
Drug: NPSP558 — 50, 75, 100 μg
  Other Names: REPEAT

SUMMARY:
This study is designed to evaluate the effect of 6-months of treatment with NPSP558 in reducing requirements for supplemental oral calcium and active vitamin D, while maintaining stable total serum calcium levels in adult subjects with hypoparathyroidism.

DETAILED DESCRIPTION:
Subjects either must have previously completed NPSP558 Study CL1-11-040 (REPLACE) including 24 weeks of active therapy and 4 weeks of follow-up to Week 28 prior to enrolling in this study or have enrolled in REPLACE and dropped out during optimization, but currently meet inclusion/exclusion criteria for REPLACE.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all the following inclusion criteria can be enrolled into this study:

1. Signed and dated informed consent form (ICF) before any study-related procedures are performed
2. Previously completed 24 weeks of therapy and 4 weeks of follow-up in the REPLACE study, OR Enrolled in REPLACE and dropped out during optimization, but currently meet inclusion/exclusion criteria for REPLACE
3. Able to perform daily SC self-injections of study medication (or have a designee perform injection) via a multidose injection pen into the thigh
4. Willingness and ability to understand and comply with the protocol
5. Women who are: (1) postmenopausal defined as 12 months amenorrhea with appropriate serum follicle stimulating hormone (FSH) levels (> 40 IU/L); (2) surgically sterilized; OR (3) of childbearing potential with a negative pregnancy test at screening and who consent to use two acceptable methods of contraception for the duration of the study, with pregnancy testing at every scheduled visit during the treatment period . Female partners (who are of childbearing potential) of male study patients must also use acceptable forms of contraception during their partner's participation

Exclusion Criteria:

Patients who meet any of the following exclusion criteria at baseline (Visit 1) are not eligible for enrollment in this study:

1. Any condition that, in the investigator's opinion after consultation with the sponsor, would preclude the safe use of NPSP558
2. Any disease or condition in the opinion of the investigator that has a high probability of precluding the patient from completing the study or where the patient cannot or will not appropriately comply with study requirements
3. Pregnant or lactating woman

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-08-19 (Actual); Primary Completion 2012-04-26 (Actual); Study Completion 2012-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (3):
- Hungary (3):
  - Semmelweis University Medical School, Budapest
  - University of Pécs, School of Medicine, Pécs
  - University of Szeged, Szeged

REFERENCES:
- [Result] Lakatos P, Bajnok L, Lagast H, Valkusz Z. AN OPEN-LABEL EXTENSION STUDY OF PARATHYROID HORMONE RHPTH(1-84) IN ADULTS WITH HYPOPARATHYROIDISM. Endocr Pract. 2016 May;22(5):523-32. doi: 10.4158/EP15936.OR. Epub 2015 Dec 18. PMID 26684150

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24 Subjects were enrolled between 8/2011 to 5/2012 at 3 Clinical sites in Hungary.
Pre-assignment Details: Subjects previously completed 24 weeks of therapy and 4 weeks of follow-up in the REPLACE study, or enrolled in REPLACE and dropped out during optimization, but currently met inclusion/exclusion criteria for REPLACE.
Groups:
- NPSP558: NPSP558: Recombinant Human Parathyroid hormone (rhPTH[1-84]) 50, 75, or 100 mcg subcutaneously daily.
Period: Overall Study
Arm/Group | NPSP558
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | NPSP558
Number analyzed (Participants) | 24
Age, Customized [Count of Participants; unit: Participants]
  < 45 years | 6
  45 to 64 years | 17
  ≥ 65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Hungary | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Achieved the Primary Triple Endpoint at Week 24, Based on Investigator Prescribed Data.
Description: A ≥ 50% reduction from baseline in dose of oral calcium or an oral calcium dose of ≤ 500 mg and a ≥ 50% reduction from baseline in dose of oral active vitamin D (calcitriol dose of ≤ 0.25 μg/day or alphacalcidol dose of ≤ 0.50 μg/day) and a total serum calcium concentration that was normalized or maintained compared to the baseline value and did not exceed the ULN of the central laboratory.
Time Frame: 24 Weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NPSP558
Number analyzed (Participants) | 24
percentage of participants | 75.0 [53.3 to 90.2]

2. Secondary Outcome: Mean Percentage Changes From Baseline in Active Vitamin D Dosages at Each Visit
Time Frame: 24 Weeks
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | NPSP558
Number analyzed (Participants) | 24
percentage of change
  Week 2 | -47.08 (31.566)
  Week 4 | -80.38 (16.688)
  Week 8 | -96.70 (7.865)
  Week 16 | -96.18 (11.521)
  Week 24 | -97.92 (10.206)

3. Secondary Outcome: Mean Percentage Changes From Baseline in Oral Calcium at Each Visit
Time Frame: 24 Weeks
Population: The Intent-to-treat population, which includes all subjects who received at least one dose of study drug and had at least one efficacy measurement.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | NPSP558
Number analyzed (Participants) | 24
percentage of change
  Week 2 | -8.3 (36.20)
  Week 4 | -46.4 (35.57)
  Week 8 | -71.5 (33.14)
  Week 16 | -71.7 (38.60)
  Week 24 | -76.0 (40.48)

4. Secondary Outcome: Proportion of Patients Achieving the Primary Endpoint at Each Visit
Description: as for outcome 1
Time Frame: 24 Weeks
Population: The Intent-to-treat population, which includes all subjects who received at least one dose of study drug and had at least one efficacy measurement .
Measure: Number; unit: percentage of participants
Arm/Group | NPSP558
Number analyzed (Participants) | 24
percentage of participants
  Week 2 | 20.8
  Week 4 | 50.0
  Week 8 | 70.8
  Week 16 | 83.3
  Week 24 | 83.3

5. Secondary Outcome: Mean Change From Baseline in 24-hour Urine Calcium Excretion
Time Frame: 24 Weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/24 hour
Arm/Group | NPSP558
Number analyzed (Participants) | 24
mg/24 hour
  Week 8 | -64.58 (188.42)
  Week 24 | -51.53 (183.41)

ADVERSE EVENTS:
Time Frame: 24 Weeks
Arm/Group | NPSP558
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 22/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NPSP558 (N=24)
Hypoaesthesia (Nervous system disorders) | 12 (23)
Headache (Nervous system disorders) | 4 (5)
Paraesthesia (Nervous system disorders) | 2 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 5 (7)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (4)
Tetany (Metabolism and nutrition disorders) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Hypoaesthesia oral (Gastrointestinal disorders) | 3 (4)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Vitamin D decreased (Investigations) | 6 (6)
Fatigue (General disorders) | 4 (6)
Polyuria (Renal and urinary disorders) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other